CLINICAL TRIAL: NCT07072429
Title: Association of Annual Hospital Volume With Mortality, Reoperation, and Length of Hospital Stay After Gastric Cancer Resection in Switzerland: A Retrospective National Registry Study
Brief Title: Annual Hospital Volume and and Short-term Postoperative Outcomes After Gastric Cancer Resection
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: Hospital volume GCR
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric cancer resection
  Interventions: Procedure: Gastric cancer resection

INTERVENTIONS:
Procedure: Gastric cancer resection — Any kind of surgical gastric cancer resection

SUMMARY:
The effect of centralisation measures on the operative outcomes after gastric cancer resection in Switzerland has not been highlighted yet. This study aims to investigate the influence of the annual hospital specific case load of gastric cancer resection on short-term postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with gastric cancer resection in Switzerland between 2013 and 2022.

Exclusion Criteria:

* incomplete case documentation
* age under 20 years
* other hospitals than general or surgical hospitals
* no index operation

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with gastric cancer resection in Switzerland between 2013 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 3112 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Periprocedural
  The association between the hospital volume and the postoperative mortality of gastric cancer resection as marginal effect with GAM (Generalized Additive Models) logistic regression

SECONDARY OUTCOMES:
Reoperation | Periprocedural
  The association between the hospital volume and the reoperation rate of gastric cancer resection as marginal effect with GAM logistic regression
Length of hospital stay | Periprocedural
  The association between the hospital volume and the length of hospital stay of gastric cancer resection as marginal effect with quantile regression.
Sociodemographic trends | 2013 - 2022

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No